CLINICAL TRIAL: NCT04360174
Title: A Prospective, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of OTX-TIC (Travoprost) Implant in Subjects With Primary Open-Angle Glaucoma or Ocular Hypertension
Brief Title: CLN-0045: Safety, and Efficacy of OTX-TIC in Participants With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-Protocol-0045
Record Dates: First submitted 2020-03-20; First posted 2020-04-24 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Sequential: Groups of participants are assigned to receive interventions based on prior milestones being reached in the study, such as in some dose escalation and adaptive design studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OTX-TIC-Cohort 1 (Experimental): 15 µg (formulation1) implant
  Interventions: Drug: OTX-TIC
- OTX-TIC-Cohort 2 (Experimental): 26 µg (formulation1) implant
  Interventions: Drug: OTX-TIC
- OTX-TIC-Cohort 3 (Experimental): 15 µg (formulation 2) implant
  Interventions: Drug: OTX-TIC
- OTX-TIC-Cohort 4 (Experimental): 5 µg (formulation 3) implant
  Interventions: Drug: OTX-TIC

INTERVENTIONS:
Drug: OTX-TIC — OTX-TIC implant is injection in the anterior chamber of the eye

SUMMARY:
To assess the safety, tolerability and efficacy of a single sustained release dose of OTX-TIC, a sustained release travoprost drug product, in subjects with primary open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open label study, to evaluate the safety, tolerability and efficacy of OTX-TIC intracameral implant in subjects with primary open-angle glaucoma or ocular hypertension. The subjects will be followed for approximately 7 months (one-month washout and 6 months follow-up after injected of the OTX-TIC implant).

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of ocular hypertension or primary open-angle glaucoma
* Have IOP that is currently controlled as assessed by the Investigator
* Have open, normal appearing anterior chamber angles as determined by gonioscopy

Exclusion Criteria:

* Have closed angle glaucoma, narrow angle glaucoma, pseudoexfoliation syndrome, pseudoexfoliation glaucoma, pigment dispersion or pigmentary glaucoma, glaucoma diagnosis prior to 15 years of age, inflammatory, neovascular or other secondary
* Have a known or suspected allergy and/or hypersensitivity to a prostaglandin (i.e. travoprost), fluorescein or to any component of the study products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Ocular Therapeutix, Inc., Petaluma, California
  - Ocular Therapeutix, Inc., Torrance, California
  - Ocular Therapeutix, Inc, Roswell, Georgia
  - Ocular Therapeutix, Inc., Austin, Texas
  - Ocular Therapeutix, Inc., Racine, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OTX-TIC-Cohort 1 | OTX-TIC-Cohort 2 | OTX-TIC-Cohort 3 | OTX-TIC-Cohort 4
Started | 5 | 4 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-TIC-Cohort 1 | OTX-TIC-Cohort 2 | OTX-TIC-Cohort 3 | OTX-TIC-Cohort 4 | Total
Number analyzed (Participants) | 5 | 4 | 5 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 2 | 2 | 5
  >=65 years | 5 | 3 | 3 | 3 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 4 | 15
  Male | 2 | 0 | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 4 | 6
  Not Hispanic or Latino | 5 | 3 | 4 | 1 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 0 | 5
  White | 5 | 2 | 2 | 5 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 5 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Ocular Treatment Emergent Adverse Events
Description: All adverse events will be captured throughout the study
Time Frame: Through study completion, 6 months
Measure: Number; unit: Number of Treatment-Emergent Events
Arm/Group | OTX-TIC-Cohort 1 | OTX-TIC-Cohort 2 | OTX-TIC-Cohort 3 | OTX-TIC-Cohort 4
Number analyzed (Participants) | 5 | 4 | 5 | 5
Number of Treatment-Emergent Events | 9 | 7 | 9 | 1

2. Primary Outcome: Efficacy Outcome
Description: IOP measurements at 8 am
Time Frame: Diurnal IOP [12 Week Visit]
Measure: Mean (Standard Deviation); unit: mmHg mean IOP change at wk12 from bln
Arm/Group | OTX-TIC-Cohort 1 | OTX-TIC-Cohort 2 | OTX-TIC-Cohort 3 | OTX-TIC-Cohort 4
Number analyzed (Participants) | 5 | 4 | 5 | 5
mmHg mean IOP change at wk12 from bln | -5.6 (2.58) | -7.0 (3.27) | -3.0 (14.4) | -7.4 (4.76)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | OTX-TIC-Cohort 1 | OTX-TIC-Cohort 2 | OTX-TIC-Cohort 3 | OTX-TIC-Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 2/4 | 3/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-TIC-Cohort 1 (N=5) | OTX-TIC-Cohort 2 (N=4) | OTX-TIC-Cohort 3 (N=5) | OTX-TIC-Cohort 4 (N=5)
Congenital, familial and genetic disorders (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Disorders (Eye disorders) | 3 (8) | 2 (7) | 2 (3) | 1 (1)
Uncoded Terms (Eye disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) — Uncoded terms in Cohort 3 consisted of 2 events of corneal edema in the Study Eye and an event of fixed and dilated pupil in the Study Eye
Investigations (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT04360174/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT04360174/SAP_001.pdf